CLINICAL TRIAL: NCT05427708
Title: Respiratory Training in the Treatment of Transdiagnostic Pathological Anxiety: A Randomized Clinical Trial
Brief Title: Respiratory Training in the Treatment of Transdiagnostic Pathological Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Freespira, Inc. (Unknown)
Responsible Party: Principal Investigator, Michael J. Telch, Professor of Psychology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002306
Record Dates: First submitted 2022-03-01; First posted 2022-06-22 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorders; Trauma; Generalized Anxiety Disorder; Panic Disorder; Agoraphobia; Illness Anxiety Disorder; Social Anxiety Disorder; Posttraumatic Stress Disorder; Acute Stress Disorder; Adjustment Disorder With Anxious Mood
Keywords: Psychoeducation; Respiratory training; Transdiagnostic; Intervention
MeSH Terms: conditions — Anxiety Disorders; Wounds and Injuries; Generalized Anxiety Disorder; Panic Disorder; Agoraphobia; Phobia, Social; Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Intervention Model Description: This study will utilize a 2 x 3 randomized controlled trial design with intervention type as a between-subjects factor with two levels (CGRI, PsyEd) and time points (baseline, posttreatment, 2-month follow-up) as a three-level within-subjects factor.
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomized by the undergraduate student coordinator for the project who is uninvolved with (1) running subjects through treatment; and (2) with data analysis. The study personnel involved in completing participants' treatment will not be blind. However, these personnel will not be involved in data maintenance or analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Capnometry-Guided Respiratory Intervention (CGRI) (Experimental): If assigned to this condition, participants will be expected to complete twice-daily 17-minute tablet-assisted breathing exercises at home for four weeks. They will also receive brief phone check-ins with their study therapist weekly to review progress and troubleshoot any problems they may be experiencing. Last, these participants will have access to a paced-breathing app that provides audio recordings to maintain specified breathing rates for up to 10 minutes.
  Interventions: Device: Capnometry-Guided Respiratory Intervention
- Psycho-Education (PsyEd) (Active Comparator): If assigned to the psycho-education condition, participants will watch pre-recorded 20-minute video presentations once-weekly for four weeks. They will meet with a study staff member to watch these videos, who will be available to answer any questions. During these sessions, they will be provided information about the nature and causes of anxiety-related disorders and learn tips for coping with anxiety symptoms when they arise. At the end of their sessions with the therapist, they will receive handouts that will help reinforce what they've learned.
  Interventions: Behavioral: Psycho-Education

INTERVENTIONS:
Device: Capnometry-Guided Respiratory Intervention — See: Arm/group descriptions
  Other Names: CGRI
  Arms: Capnometry-Guided Respiratory Intervention (CGRI)
Behavioral: Psycho-Education — See: Arm/group descriptions
  Other Names: PsyEd
  Arms: Psycho-Education (PsyEd)

SUMMARY:
Purpose of the Research: The primary aim of the proposed study is to conduct a randomized parallel-group 2-arm clinical trial investigating capnometry-guided respiratory intervention (CGRI) for pathological anxiety. CGRI aims to raise end-tidal CO2 levels thereby lowering hyperventilation-induced respiratory alkalosis and its associated fear-eliciting somatic reactions. Psycho-education about anxiety and its effects (PsyEd) will serve as a credible control comparator.

DETAILED DESCRIPTION:
Low end-tidal CO2 (ETCO2), which is an accompanying feature of hyperventilation, has been associated with a variety of anxiety disorders, including panic disorder and social phobia. More recently, researchers have examined the efficacy of capnometry-guided respiratory intervention (CGRI) as a method for increasing ETCO2 and thereby reducing hyperventilation-induced anxiety/panic symptoms. Promising preliminary efficacy studies have shown that CGRI results in decreased panic symptom frequency and severity at a rate comparable to that of cognitive therapy. A recent uncontrolled proof-of-concept study showed that CGRI led to significant reductions in trauma symptoms in a sample of patients meeting DSM-5 criteria for PTSD. However, CGRI has not been adequately evaluated in the treatment of anxiety disorders other than panic disorder with or without agoraphobia.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically elevated anxiety as indicated by an eight or higher on the Overall Anxiety Severity and Impairment Scale (OASIS).
2. Meets DSM-5 criteria for one or more of the following anxiety or trauma-related disorders as their "primary" mental disorder:

   * Generalized Anxiety Disorder
   * Panic Disorder
   * Health Anxiety
   * Agoraphobia
   * Social Anxiety Disorder
   * Posttraumatic Stress Disorder
   * Acute Stress Disorder
   * Adjustment Disorder with primary anxious mood
   * Anxiety disorder not otherwise specified
3. No current use of psychotropic medications or stable on current medications for at least 6 weeks
4. Age 18+.
5. Able to arrange transportation to our laboratory for study appointments.
6. Fluent in English.

Exclusion Criteria:

1. No history of medical conditions that would contraindicate participation in fear-provocation or respiratory challenges, including:

   * Cardiovascular or respiratory disorders
   * High blood pressure
   * Epilepsy
   * Strokes
   * Seizures
   * History of fainting
   * Pregnant or lactating
2. Not currently receiving other psychological treatment for anxiety.
3. No history of a suicide attempt within the past 6 months.
4. No history of psychosis within the past 6 months.
5. No history of moderate to severe alcohol or substance use disorder (with the exception of nicotine) within the past 3 months.
6. Does not endorse COVID-19 symptoms during the screening phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale | Pre-Treatment (Week 0), Post-treatment (Week 5), 2-Month Follow-Up (Week 13)
  Change from baseline in self-reported transdiagnostic anxiety symptoms (range = 0 - 20, with higher scores indexing more symptoms).
Computerized Hamilton Anxiety Scale | Pre-Treatment (Week 0), Post-treatment (Week 5), 2-Month Follow-Up (Week 13)
  Change from baseline in anxiety symptom severity. Each item is assessed both in terms of frequency and severity. Scores on these probes are summed and divided by the number of response options. Higher scores index higher severity.

SECONDARY OUTCOMES:
Sheehan Disability Scale | Pre-Treatment (Week 0), Weekly Assessments (Weeks 1 - 4), Post-treatment (Week 5), 2-Month Follow-Up (Week 13)
  Change from baseline in overall disability (range = 0 - 30, with higher scores indexing more disability).
PROMIS - Global Health (Mental Health Subdomain) | Pre-Treatment (Week 0), Weekly Assessments (Weeks 1 - 4), Post-treatment (Week 5), 2-Month Follow-Up (Week 13)
  Change from baseline in quality of life (range = 4 - 20, with higher scores indexing higher quality of life).
Anxiety Sensitivity Composite Measure | Pre-Treatment (Week 0), Weekly Assessments (Weeks 1 - 4), Post-treatment (Week 5), 2-Month Follow-Up (Week 13)
  This composite measure will incorporate scores on the Anxiety Sensitivity Index-3 (ASI-3), Body Sensations Questionnaire (BSQ), and Texas Multi-Factor Anxiety Sensitivity Scale (TMASS). Scores on each of these individual measures will be transformed into z scores and then averaged to derive this composite index. We will measure change from baseline in anxiety sensitivity.
Modified DIAMOND | Pre-Treatment (Week 0), 2-Month Follow-Up (Week 13)
  Change from baseline in DIAMOND Diagnostic Interview + Health Anxiety Questionnaire scores.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reiss S, Peterson RA, Gursky DM, McNally RJ. Anxiety sensitivity, anxiety frequency and the prediction of fearfulness. Behav Res Ther. 1986;24(1):1-8. doi: 10.1016/0005-7967(86)90143-9. No abstract available. PMID 3947307
- [Background] Li W, Zinbarg RE. Anxiety sensitivity and panic attacks: a 1-year longitudinal study. Behav Modif. 2007 Mar;31(2):145-61. doi: 10.1177/0145445506296969. PMID 17307932
- [Background] Maller RG, Reiss S. Anxiety sensitivity in 1984 and panic attacks in 1987. J Anxiety Disord. 1992;6(3):241-247.
- [Background] Schmidt NB, Lerew DR, Jackson RJ. Prospective evaluation of anxiety sensitivity in the pathogenesis of panic: replication and extension. J Abnorm Psychol. 1999 Aug;108(3):532-7. doi: 10.1037//0021-843x.108.3.532. PMID 10466277
- [Background] Telch MJ, Rosenfield D, Lee HJ, Pai A. Emotional reactivity to a single inhalation of 35% carbon dioxide and its association with later symptoms of posttraumatic stress disorder and anxiety in soldiers deployed to Iraq. Arch Gen Psychiatry. 2012 Nov;69(11):1161-8. doi: 10.1001/archgenpsychiatry.2012.8. PMID 23117637
- [Background] Cobb AR, Lancaster CL, Meyer EC, Lee HJ, Telch MJ. Pre-deployment trait anxiety, anxiety sensitivity and experiential avoidance predict war-zone stress-evoked psychopathology. Journal of Contextual Behavioral Science. 2017;6(3):276-287.
- [Background] Schmidt NB, Telch MJ. Role of fear of fear and safety information in moderating the effects of voluntary hyperventilation. Behav Ther. 1994;25(2):197-208.
- [Background] Beck JG, Shipherd JC, Zebb BJ. How does interoceptive exposure for panic disorder work? An uncontrolled case study. J Anxiety Disord. 1997 Sep-Oct;11(5):541-56. doi: 10.1016/s0887-6185(97)00030-3. PMID 9407272
- [Background] Craske MG, Barlow DH. Mastery of Your Anxiety and Panic: Therapist Guide. Published online 2006. doi:10.1093/med:psych/9780195311402.001.0001
- [Background] Margraf J, Barlow DH, Clark DM, Telch MJ. Psychological treatment of panic: work in progress on outcome, active ingredients, and follow-up. Behav Res Ther. 1993 Jan;31(1):1-8. doi: 10.1016/0005-7967(93)90036-t. PMID 8093337
- [Background] Telch MJ, Lucas JA, Schmidt NB, Hanna HH, LaNae Jaimez T, Lucas RA. Group cognitive-behavioral treatment of panic disorder. Behav Res Ther. 1993 Mar;31(3):279-87. doi: 10.1016/0005-7967(93)90026-q. PMID 8476402
- [Background] Ley R. Blood, breath, and fears: A hyperventilation theory of panic attacks and agoraphobia. Clin Psychol Rev. 1985;5(4):271-285.
- [Background] Studer RK, Danuser B, Hildebrandt H, Arial M, Wild P, Gomez P. Hyperventilation in anticipatory music performance anxiety. Psychosom Med. 2012 Sep;74(7):773-82. doi: 10.1097/PSY.0b013e31825e3578. Epub 2012 Jul 23. PMID 22826290
- [Background] Kaplan A, Mannarino AP, Nickell PV. Evaluating the Impact of Freespira on Panic Disorder Patients' Health Outcomes and Healthcare Costs within the Allegheny Health Network. Appl Psychophysiol Biofeedback. 2020 Sep;45(3):175-181. doi: 10.1007/s10484-020-09465-0. PMID 32342249
- [Background] Meuret AE, Wilhelm FH, Ritz T, Roth WT. Feedback of end-tidal pCO2 as a therapeutic approach for panic disorder. J Psychiatr Res. 2008 Jun;42(7):560-8. doi: 10.1016/j.jpsychires.2007.06.005. Epub 2007 Aug 3. PMID 17681544
- [Background] Tolin DF, McGrath PB, Hale LR, Weiner DN, Gueorguieva R. A Multisite Benchmarking Trial of Capnometry Guided Respiratory Intervention for Panic Disorder in Naturalistic Treatment Settings. Appl Psychophysiol Biofeedback. 2017 Mar;42(1):51-58. doi: 10.1007/s10484-017-9354-4. PMID 28194546
- [Background] Meuret AE, Rosenfield D, Seidel A, Bhaskara L, Hofmann SG. Respiratory and cognitive mediators of treatment change in panic disorder: evidence for intervention specificity. J Consult Clin Psychol. 2010 Oct;78(5):691-704. doi: 10.1037/a0019552. PMID 20873904
- [Background] Ostacher MJ, Fischer E, Bowen ER, Lyu J, Robbins DJ, Suppes T. Investigation of a Capnometry Guided Respiratory Intervention in the Treatment of Posttraumatic Stress Disorder. Appl Psychophysiol Biofeedback. 2021 Dec;46(4):367-376. doi: 10.1007/s10484-021-09521-3. PMID 34468913